CLINICAL TRIAL: NCT05578625
Title: Circulating Tumor DNA Methylation Sequencing for Multiple Myeloma Minimal Residual Disease Detection and Clonal Evolution Monitoring
Brief Title: ctDNA Methylation Sequencing for Myeloma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Collaborators: MethylGene Tech Co., Ltd. China (Unknown)
Responsible Party: Principal Investigator, Gang An, Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Science & Peking Union Medical College, Institute of Hematology & Blood Diseases Hospital, China
Other Study IDs: ctDNA-MM-2022
Record Dates: First submitted 2022-09-07; First posted 2022-10-13 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Multiple Myeloma
Keywords: circulationg tumor DNA; methylation sequencing; minimal residual disease; clonal evolution
MeSH Terms: conditions — Multiple Myeloma; Neoplasm, Residual

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Myeloma: This study includes a total of 60 multiple myeloma patients, and peripheral blood will be collected at newly diagnosed, remission after 4 cycles of therapy, and, relapse stage.
  Interventions: Other: plasma circulation DNA methylation sequencing

INTERVENTIONS:
Other: plasma circulation DNA methylation sequencing — 10 mL of peripheral blood will be drawn from 60 multiple myeloma patients at diagnosis, 4 months post-induction, and at relapse, and cell-free DNA is then extracted and undergo bisulfite methylation sequencing.

SUMMARY:
1. To carry out research on minimal residual disease (MRD) monitoring in patients with multiple myeloma (MM) based on plasma circulating tumor DNA (ctDNA) methylation sequencing, which aims to explore new MRD detection methods for MM;
2. Carry out ctDNA-based methylation sequencing in newly diagnosed, remission, and, relapsed MM patients, to track the clonal evolution patterns; and explore the in the initial diagnosis-remission-relapse stage of MM, track the clonal evolution characteristics of methylation profiles in MM patients during the disease progression.

ELIGIBILITY:
Inclusion Criteria:

- For myeloma patients: i) Age no less than 18 and no more than 75; ii) Diagnosed with symptomatic multiple myeloma according to IMWG consensus; iii) Provide informed consent in accordance with the declaration of Helsinki.

- For healthy controls: i) Age no less than 18 and no more than 75; ii) Provide informed consent in accordance with the declaration of Helsinki.

Exclusion Criteria:

- For myeloma patients: i) Insufficient amount of peripheral blood obtained; ii) Methylation sequencing failed due to technical reasons.

- For healthy controls: i) Insufficient amount of peripheral blood obtained; ii) Methylation sequencing failed due to technical reasons.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: For patients aged between 18 and 75, and diagnosed with symptomatic multiple myeloma according to IMWG consensus will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Sample Collection Completed | From Aug 31 2022 to Jun 30 2025
  When the peripheral blood samples required for the study have been collected

CONTACTS AND LOCATIONS:
Overall Officials: InsituteHBDH, Principal Investigator — Institute of Hematology and Blood Diseases Hospital,Tianjin, China, 300020
Locations (1):
- Institute of Hematology and Blood Diseases Hospital Chinese Academy of Medical Sciences, Tianjin, China

IPD SHARING:
Plan to Share IPD: No
The datasets generated during and/or analysed during the current study are available from the corresponding author at angang@ihcams.ac.cn on reasonable request.